CLINICAL TRIAL: NCT00609128
Title: Expression of Inflammatory Mediators in Allergic Conjunctivitis
Brief Title: Effect of Olopatadine on Allergic Tear Mediators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1998-381; R01EY012526 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-02-06 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Allergic Conjunctivitis
Keywords: tears; conjunctival epithelial cells; olopatadine; eosinophils
MeSH Terms: conditions — Conjunctivitis, Allergic; Lacerations | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olopatadine (Experimental): one drop in one eye only two times per day at an interval of 6 to 8 hours for 1 week
  Interventions: Drug: olopatadine

INTERVENTIONS:
Drug: olopatadine — olopatadine one drop in one eye for one week

SUMMARY:
The purpose of the research is to determine which inflammatory substances are involved in causing allergic symptoms in the eye. Allergic conjunctivitis is a common problem with symptoms of temporary redness, itching, tearing, and swelling of the eyes. Substances released by cells in the affected tissues cause allergic reactions in the eye and elsewhere in the body.

DETAILED DESCRIPTION:
Ocular allergies are extremely common, affecting up to 80 million people in the USA. Our research question is:

Are there differences in inflammatory mediators and cell surface activation markers in patients undergoing seasonal allergic conjunctivitis compared to those with sight threatening disease such as Atopic Keratoconjunctivitis (AKC) and will the use of the anti-allergy eye drop, PATANOL® (olopatadine hydrochloride) affect these parameters?

Experimental Design:

Ocular surface cells (by impression cytology) and tears (via capillary tube) are collected from allergic, non-allergic, and AKC subjects undergoing an reaction induced either by seasonal allergen or topical allergen provocation (specificity and dose determined via skin testing). Ocular surface cells are evaluated for surface activation markers. Tears are evaluated for mediator content. Tears are also incubated with peripheral blood eosinophils and lymphocytes to see effects on adhesion to conjunctival epithelial cells.

ELIGIBILITY:
Inclusion Criteria:

* Skin test positive
* Able to put drops in eyes
* Able to have tears collected

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal P Barney, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Background] Cook EB. Tear cytokines in acute and chronic ocular allergic inflammation. Curr Opin Allergy Clin Immunol. 2004 Oct;4(5):441-5. doi: 10.1097/00130832-200410000-00018. PMID 15349046
- [Result] Cook EB, Stahl JL, Brooks AM, Graziano FM, Barney NP. Allergic tears promote upregulation of eosinophil adhesion to conjunctival epithelial cells in an ex vivo model: inhibition with olopatadine treatment. Invest Ophthalmol Vis Sci. 2006 Aug;47(8):3423-9. doi: 10.1167/iovs.06-0088. PMID 16877412

RESULTS

PARTICIPANT FLOW:
Groups:
- Olopatadine: one drop olopatadine in one eye only, two times per day at an interval of 6 to 8 hours for 1 week. This allows the untreated eye to be the control.
Period: Overall Study
Arm/Group | Olopatadine
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Olopatadine Treatment (Only One Eye): one drop olopatadine in one eye only, two times per day at an interval of 6 to 8 hours for 1 week. This allows the untreated eye to be the control.
Arm/Group | Olopatadine Treatment (Only One Eye)
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 8
Region of Enrollment [Number; unit: participants] — tears were collected from olopatadine treated eye and untreated eye of participants . tears were collected from 21 participants ( not 42) not all collected tears were used in final experiments.
  participants
    United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Study Examined Whether the Incubation of Human Conjunctival Epithelial Cells With Tears Pooled From Allergic Subjects (One Eye With and Other Eye Without Olopatadine Treatment) Promotes Eosinophil Adhesion
Description: Outcome:
  The collected tears (from 10 subjects)were pooled, incubated with primary conjunctival epithelial cells before eosinophil adhesion was measured via eosinophil peroxidase assay.
  Eosinophils in eosinophils / square cm measured.
Time Frame: 1 week for tear collection, tears stored at - 80 C until used
Measure: Mean (Standard Error); unit: eosinophils/square cm epithelial cells
Groups:
- Tears From Olopatadine Treated Eyes; Tears From Untreated Eyes: Allergic subjects treated one eye with olopatadine and did not treat other eye (control). Tears collected from both eyes and incubated with conjunctival epithelial cells. We determined whether tears collected from olopatadine treated eyes of subjects result in more or less purified peripheral blood eosinophil adhesion to conjunctival epithelial cells compared to tears collected from untreated eyes from the same subjects.
Arm/Group | Tears From Olopatadine Treated Eyes | Tears From Untreated Eyes
Number analyzed (Participants) | 10 | 10
eosinophils/square cm epithelial cells | 4517 (485) | 5004 (445)
Statistical Analysis 1: Comparison: Tears From Olopatadine Treated Eyes; tears were collected in season from eyes of allergic patients with or without olopatadine treatment, that is one eye was treated and the patients other eye was not. Tears from each patient's eyes were pooled to provide enough volume; Test type: Superiority or Other; p < 0.05, ANOVA; ANOVA with preplanned comparisons was used to generate two tailed P values. Paired t tests were used to make appropriate post-ANOVA comparisons

ADVERSE EVENTS:
Arm/Group | Olopatadine
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No